CLINICAL TRIAL: NCT01980316
Title: Phase 4 Study of Argatroban for Preventing Restenosis After Extracranial Vertebral Artery Stenting
Brief Title: Argatroban for Preventing Occlusion and Restenosis After Extracranial Vertebral Artery Stenting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xinfeng Liu (Other)
Responsible Party: Sponsor-Investigator, Xinfeng Liu, Argatroban for Preventing Restenosis After Extracranial vertebral Artery Stenting, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JLH3
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: CVD
Keywords: Argatroban; Extracranial vertebral Artery Stenting; restenosis
MeSH Terms: interventions — argatroban; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Argatroban group (Experimental): Argatroban in patients undergoing load 250μg/kg, followed by 15μg/kg/min continuous intravenous infusion.5 days after surgery, take 10mg intravenous infusion of speed 2/day
  Interventions: Drug: Argatroban; Drug: non-argatroban treated group
- non-argatroban treated group (Experimental): Patients in control group will receive Unfractionated heparin treatment
  Interventions: Drug: Argatroban; Drug: non-argatroban treated group

INTERVENTIONS:
Drug: Argatroban — Argatroban in patients undergoing load 250μg/kg, followed by 15μg/kg/min continuous intravenous infusion.5 days after surgery, take 10mg intravenous infusion of speed 2/day
Drug: non-argatroban treated group — Patients in control group will receive Unfractionated heparin treatment
  Other Names: Unfractionated heparin

SUMMARY:
Argatroban is a selective thrombin inhibitor, and previous study had suggested that argatroban use post percutaneous coronary intervention could potentially prevent reocclusion. But there has no study on large sample of argatroban treated restenosis vertebral artery stenting. This study will test the safety and efficacy of the argatroban on prevent Occlusion and Restenosis in patients with Extracranial vertebral Artery Stenting.

DETAILED DESCRIPTION:
The risk of restenosis post intracranial and extracranial artery stenting is 20-40%, therefore, in the past, aspirin and clopidogrel were performed as anticoagulant therapy post stenting.But this treatment had limited effectiveness upon restenosis. Argatroban is a selective thrombin inhibitor, and previous study had suggested that argatroban use post PCI could potentially prevent reocclusion. But there has no study on large sample of argatroban treated Occlusion and Restenosis Extracranial vertebral Artery Stenting. This study will test the safety and efficacy of the argatroban on prevent Occlusion and Restenosis in patients with Extracranial vertebral Artery Stenting.

ELIGIBILITY:
Inclusion Criteria:

* For Extracranial vertebral Artery lesion, stenting was considered for symptomatic stenosis≥50% or asymptomatic stenosis≥70%;
* Successfully had intracranial or extracranial artery stenting.

Exclusion Criteria:

* Evidence of hemorrhagic brain infarction, intracranial and extracranial hematoma, or intraventricular hemorrhage, or Gastrointestinal ulcers in 3 months
* Hypersensitivity to contrast agent
* Malignant hypertension
* Difficult to perform the vertebral artery stenting
* Severe hepatic or cardiac disorders, infectious disorders, dehydration, etc.
* Difficult to hand follow-up visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
restenosis | at half a year
  Stenosis detected by DSA(digital subtraction angiography),CTA(CT angiography)or MRA(MR angiography)was measured according to NASCET(North American Symptomatic Carotid Endarterectomy Trial)method.Concretely, NASCET stenosis is calculated from the ratio of the linear luminal diameter of the narrowest segment of the diseased portion of the artery to the diameter of the artery beyond any poststenotic dilatation: NASCET=(1-md/C)×100%

SECONDARY OUTCOMES:
NIHSS, mRS | at half a year
  NIHSS and mRS are widely used stroke deficit assessment tools. Most clinical stroke-related trials require a baseline and outcome severity assessment. The baseline of mRS is rank 0, NIHSS 0; the severity of mRS is 6, NIHSS 42. AS many patients have one or more strokes before they perform stenting, this study selected NIHSS and mRS as the supplementary materials to estimate the stroke deficit of patients and to reflect the therapeutic effect and safety of stenting and argatroban therapy. These two scales are performed according to the guidance before and after stenting and argatroban therapy.

OTHER OUTCOMES:
Various adverse effects | at half a year

CONTACTS AND LOCATIONS:
Overall Officials: Xinfeng Liu, MD, Study Chair — Department of Neurology, Jinling Hospital, Nanjing University School of Medicine
Locations (1):
- Department of Neurology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu, China